CLINICAL TRIAL: NCT03392285
Title: Undisplaced Femoral Neck Fractures: Treatment With Internal Fixation or Hip Arthroplasty
Brief Title: Undisplaced Femoral Neck Fractures
Acronym: UNFNF
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UFNF_IFvsHA
Record Dates: First submitted 2018-01-01; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Hip Fractures; Femoral Neck Fractures; Undisplaced Fracture; Internal Fixation; Complications; Arthroplasty Complications
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Internal fixation: Patients above 65years old with an undisplaced femoral neck fractures treated with primary internal fixation with screws.
  Interventions: Device: Internal fixation or hip arthroplasty
- Hip arthroplasty: Patients above 65years old with a displaced femoral neck fractures treated with primary hip arthroplasty.
  Interventions: Device: Internal fixation or hip arthroplasty

INTERVENTIONS:
Device: Internal fixation or hip arthroplasty — Patients treated according to the routine at the orthopedic department with screw fixation of an undisplayed femoral neck fracture or hip arthroplasty for a displaced femoral neck fracture.

SUMMARY:
Purpose The purpose of this study is to compare the clinical outcome and the rate of reoperations in a cohort of patients with undisplaced femoral neck fractures treated with internal fixation and patients with displaced femoral neck fractures treated with hip arthroplasty.

Methods In a consecutive series of patients we compared the results of internal fixation for undisplaced femoral neck fractures with those of hip arthroplasty for displaced fractures (control group) of elderly patients. Risk of reoperation and patient reported hip function assessed with Harris hip score and WOMAC were used as outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

Above 65 years old Displaced femoral neck fracture treated with hip arthroplasty Undisplaced femoral neck fracture treated with internal fixation

Exclusion Criteria:

* Pathologic fracture

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: To evaluate the potential benefit of surgery with arthroplasty. All patients treated at Sundsvall hospital, Sweden for a displaced femoral neck fracture treated with hip arthroplasty or a undisplaced femoral neck fracture treated with internal fixation were included in a prospective cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Reoperation | 4 years
  Reapportions are recorded and compared between the groups.

SECONDARY OUTCOMES:
Harris hip score | 1 year postoperatively
  Patient reported outcome (0-100 points) for evaluation of hip function.
WOMAC | 1 year postoperatively
  Patient reported outcome (0-96 points) for evaluation of hip function.
Pain in the operated hip | 1 year postoperatively
  Estimated with pain numeric rating scale (PNRS). Grading 0-10.

IPD SHARING:
Plan to Share IPD: No
If researchers requests data - anonymous data will be shared.

REFERENCES:
- [Background] Rogmark C, Flensburg L, Fredin H. Undisplaced femoral neck fractures--no problems? A consecutive study of 224 patients treated with internal fixation. Injury. 2009 Mar;40(3):274-6. doi: 10.1016/j.injury.2008.05.023. Epub 2008 Dec 13. PMID 19070851
- [Background] Gjertsen JE, Dybvik E, Furnes O, Fevang JM, Havelin LI, Matre K, Engesaeter LB. Improved outcome after hip fracture surgery in Norway. Acta Orthop. 2017 Oct;88(5):505-511. doi: 10.1080/17453674.2017.1344456. Epub 2017 Jul 6. PMID 28681677
- [Background] Han SK, Song HS, Kim R, Kang SH. Clinical results of treatment of garden type 1 and 2 femoral neck fractures in patients over 70-year old. Eur J Trauma Emerg Surg. 2016 Apr;42(2):191-6. doi: 10.1007/s00068-015-0528-6. Epub 2015 Apr 18. PMID 26038046
- [Background] Chen WC, Yu SW, Tseng IC, Su JY, Tu YK, Chen WJ. Treatment of undisplaced femoral neck fractures in the elderly. J Trauma. 2005 May;58(5):1035-9; discussion 1039. doi: 10.1097/01.ta.0000169292.83048.17. PMID 15920421
- [Background] Gjertsen JE, Fevang JM, Matre K, Vinje T, Engesaeter LB. Clinical outcome after undisplaced femoral neck fractures. Acta Orthop. 2011 Jun;82(3):268-74. doi: 10.3109/17453674.2011.588857. PMID 21619501
- [Derived] Mukka S, Sjoholm P, Aziz A, Eisler T, Kadum B, Krupic F, Morberg P, Sayed-Noor A. A cohort study comparing internal fixation for undisplaced versus hip arthroplasty for displaced femoral neck fracture in the elderly: a pilot study for a clinical trial. Pilot Feasibility Stud. 2020 Jul 11;6:98. doi: 10.1186/s40814-020-00642-w. eCollection 2020. PMID 32670600